CLINICAL TRIAL: NCT01094054
Title: Adjustable Gastric Banding and Its Effects on Postprandial Glucose Metabolism Independent of Weight Loss
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Adrian Vella, Professor of Medicine, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 09-008460
Record Dates: First submitted 2010-03-24; First posted 2010-03-26 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Obesity; Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary and lifestyle modification (Active Comparator): Patients in this arm will eat meals that are identical in size and caloric composition to those consumed by participants in the other arm who undergo adjustable gastric banding
  Interventions: Behavioral: Dietary and lifestyle modification
- Adjustable gastric banding (Experimental): Subjects will undergo gastric banding as per clinical practice
  Interventions: Procedure: Adjustable gastric banding

INTERVENTIONS:
Procedure: Adjustable gastric banding — Placement of adjustable gastric band - laparoscopically
  Arms: Adjustable gastric banding
Behavioral: Dietary and lifestyle modification — Dietary and lifestyle modification
  Subjects will meet with a dietitian and a psychologist on a weekly basis and consume a diet matched to that of the banding arm
  Arms: Dietary and lifestyle modification

SUMMARY:
The overall aim is to determine the mechanism(s) by which common bariatric surgical procedures alter carbohydrate metabolism. Understanding these mechanisms may ultimately lead to the development of novel interventions for the prevention and treatment of Type 2 diabetes and obesity.

DETAILED DESCRIPTION:
The overall aim of this application is to determine the mechanism(s) by which common bariatric surgical procedures alter carbohydrate metabolism. Very often, resolution of diabetes occurs in the early post-operative period prior to the development of significant weight loss. It has been suggested that bariatric surgery alters insulin action but few studies have examined insulin secretion or postprandial glucose fluxes in such patients. At the present time, little is known about how the various bariatric surgical procedures alter glucose homeostasis. It is essential that the effect of bariatric surgery and meal size on these parameters be understood and accurately measured. Enteroendocrine secretion is affected by the rate of intestinal delivery of calories and may also be modulated by the enteric nervous system and the rate of direct delivery of nutrients to enteroendocrine cells. Direct measurement of intestinal transit is also an important part of understanding how bariatric surgery alters intestinal secretion of hormones that may alter glucose metabolism. The Oral and C-peptide Minimal Models when applied to C-peptide, glucose and insulin concentrations after ingestion of a standard labeled mixed meal can accurately measure insulin secretion and action. Subsequently, the disposition index provides a measurement of the appropriateness of insulin secretion for the prevailing insulin action. When coupled with established triple-tracer methodology, a mixed meal can be used to measure fasting and postprandial glucose fluxes. The present experiments will determine the mechanism of glucose lowering after adjustable gastric banding (AGB). AGB seems to be superior to medical therapy in type 2 diabetes. However, bariatric surgery was not compared to intensive efforts at weight reduction which itself ameliorates diabetes and cardiovascular risk. It is therefore unknown if the beneficial effects of AGB on glucose metabolism are related to weight-loss per se rather than a direct effect of AGB.

ELIGIBILITY:
* Individuals aged 30 - 65 years seen in the Nutrition Clinic at the Mayo Clinic, are potentially eligible prior to undergoing adjustable gastric banding (AGB).
* We will recruit 20 subjects who have a fasting glucose concentration of 126 mg/dl on two or more occasions or who have a history of type 2 diabetes treated with one or two oral agents other than thiazolidinediones.
* Potential participants will attend the Mayo Clinic Clinical Research Unit (CRU) for a screening visit.
* In addition, the investigators will also recruit 20 subjects with type 2 diabetes, from the Nutrition Clinic who are not interested in pursuing surgical intervention.
* The 2 groups will be matched for age, gender and BMI and duration and severity (HbA1c and no. of oral medications needed to achieve glycemic control) of diabetes.

Exclusion Criteria:

* Subjects less than 30 years of age or who are on insulin will not be studied to minimize the possibility of type 1 diabetes.
* Subjects older than 65 years of age will not be studied to minimize the potential confounding effects of age on glucose tolerance.
* Healthy status will indicate that the participant has no known active systemic illness and no history of microvascular or macrovascular complications of their diabetes.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Disposition Index | Change compared to baseline 12 weeks after intervention
  Insulin sensitivity which measures the overall ability of insulin to stimulate glucose disposal and inhibit glucose production will be calculated from plasma glucose and insulin concentrations using the "oral" glucose minimal model. Beta-cell responsivity indices will be calculated using plasma glucose and C-peptide concentrations using the oral C-peptide minimal model. The appropriateness of insulin secretion for the prevailing degree of insulin action is assessed by calculating the total disposition index (DItotal), which equals the product of insulin secretion and insulin sensitivity.

SECONDARY OUTCOMES:
Gastric emptying and intestinal transit | change compared to baseline 12 weeks after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Sathananthan M, Shah M, Edens KL, Grothe KB, Piccinini F, Farrugia LP, Micheletto F, Man CD, Cobelli C, Rizza RA, Camilleri M, Vella A. Six and 12 Weeks of Caloric Restriction Increases beta Cell Function and Lowers Fasting and Postprandial Glucose Concentrations in People with Type 2 Diabetes. J Nutr. 2015 Sep;145(9):2046-51. doi: 10.3945/jn.115.210617. Epub 2015 Aug 5. PMID 26246321